CLINICAL TRIAL: NCT06249698
Title: Impact of Active Nutrition Program on Weight Loss and Associated Measures of Health in Overweight and Obese Men and Women
Brief Title: Active Nutrition Program on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: USANA Health Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO-FY2022-181
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Weight Loss
Keywords: Active Nutrition
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Experimental randomly assigned unblinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Nutrition program (Experimental): Subjects in this arm will follow the Active Nutrition program for 60 days with study visits at 0 days, 30 days, and 60 days.
  Interventions: Dietary Supplement: meal replacements and supplements
- Regular Diet (No Intervention): Subjects in this arm will follow their regular diet for 60 days with study visits at 0 days, 30 days, and 60 days.

INTERVENTIONS:
Dietary Supplement: meal replacements and supplements — Consumed daily: 2 Nutrimeal Active meal replacement shake, 1 electrolyte replacement drink, 3 metabolism + supplements, 1 whole food meal, and whole food snacks consisting of fruits and vegetables. 1200-1600 calories per day
  Arms: Active Nutrition program

SUMMARY:
The study will evaluate the impact of the Active Nutrition 60-day program from USANA on weight loss and related measures, such as body composition, physical appearance/body shape, perceived wellness, and biochemical markers of health (e.g., blood lipids, glucose, insulin).

DETAILED DESCRIPTION:
To date, no controlled study exists to evaluate the impact of the Active Nutrition program from USANA on weight loss and related measures, such as body composition, physical appearance/body shape, perceived wellness, and biochemical markers of health (e.g., blood lipids, glucose, insulin). Therefore, the purpose of the proposed study is to evaluate the Active Nutrition weight loss program on body weight and related variables in a sample of overweight and obese men and women. Subjects in the Active Nutrition group will be compared to a control group of men and women following their standard diet, for a period of 60 days.

ELIGIBILITY:
Inclusion Criteria:

* body mass index 28-39.9 kilograms per square meter
* weigh less than 500 lbs
* able to fast overnight (greater than 10 hours)

Exclusion Criteria:

* tobacco user
* diagnosed with type 1 or 2 diabetes
* diagnosed with liver disease
* adversity to fiber or protein supplements
* allergic to any of the ingredients
* taking a weight loss dietary supplement or adhering to a weight loss plan for the month prior to or during the study
* consumption of alcohol within 24 hours of study visit
* consumption of caffeine within 24 hours of study visit
* strenuous exercise within 24 hours of study visit
* self-reported active infection or illness
* pregnant or lactating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-08-19 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Lipids | 0 days of assigned diet (baseline)
  Blood lipids (cholesterol, high density lipids, low density lipids, triglycerides and very low density lipids) will be measured in milligram per deciliter (mg/dL).
Lipids | 30 days of assigned diet
  Blood lipids (cholesterol, high density lipids, low density lipids, triglycerides and very low density lipids) will be measured in mg/dL.
Lipids | 60 days of assigned diet
  Blood lipids (cholesterol, high density lipids, low density lipids, triglycerides and very low density lipids) will be measured in mg/dL.
Glucose | 0 days of assigned diet (baseline)
  Glucose will be measured in whole blood using a glucometer in mg/dL.
Glucose | 30 days of assigned diet
  Glucose will be measured in whole blood using a glucometer in mg/dL.
Glucose | 60 days of assigned diet
  Glucose will be measured in whole blood using a glucometer in mg/dL.
Insulin | 0 days of assigned diet (baseline)
  Insulin will be measured from serum in micro-international units per milliliter.
Insulin | 30 days of assigned diet
  Insulin will be measured from serum in micro-international units per milliliter.
Insulin | 60 days of assigned diet
  Insulin will be measured from serum in micro-international units per milliliter.
Body Weight | 0 days of assigned diet (baseline)
  Body weight will determined in kilograms using a digital scale.
Body Weight | 30 days of assigned diet
  Body weight will determined in kilograms using a digital scale.
Body Weight | 60 days of assigned diet
  Body weight will determined in kilograms using a digital scale.
Waist circumference | 0 days of assigned diet (baseline)
  Waist circumference will be measured in centimeter.
Waist circumference | 30 days of assigned diet
  Waist circumference will be measured in centimeter.
Waist circumference | 60 days of assigned diet
  Waist circumference will be measured in centimeter.
Hip circumference | 0 days of assigned diet (baseline)
  Hip circumference will be measured in centimeter.
Hip circumference | 30 days of assigned diet
  Hip circumference will be measured in centimeter.
Hip circumference | 60 days of assigned diet
  Hip circumference will be measured in centimeter.
Body Mass Index | 0 days of assigned diet (baseline)
  body mass index will be calculated in kg per square meter from height and weight measurements.
Body Mass Index | 30 days of assigned diet
  body mass index will be calculated in kg per square meter from height and weight measurements.
Body Mass Index | 60 days of assigned diet
  body mass index will be calculated in kg per square meter from height and weight measurements.
Body composition percentages | 0 days of assigned diet (baseline)
  body composition percentages of fat and lean mass will be determined via Dual-energy x-ray absorptiometry.
Body composition percentages | 30 days of assigned diet
  body composition percentages of fat and lean mass will be determined via Dual-energy x-ray absorptiometry.
Body composition percentages | 60 days of assigned diet
  body composition percentages of fat and lean mass will be determined via Dual-energy x-ray absorptiometry.
Body composition mass | 0 days of assigned diet (baseline)
  Body composition masses of fat, lean mass, visceral fat, and bone mineral in grams will be determined via Dual-energy x-ray absorptiometry.
Body composition mass | 30 days of assigned diet
  Body composition masses of fat, lean mass, visceral fat, and bone mineral in grams will be determined via Dual-energy x-ray absorptiometry.
Body composition mass | 60 days of assigned diet
  Body composition masses of fat, lean mass, visceral fat, and bone mineral in grams will be determined via Dual-energy x-ray absorptiometry.
Resting Heart Rate | 0 days of assigned diet (baseline)
  Heart Rate will be determined in beats per minute using an automated blood pressure cuff following a 10 minute rest.
Resting Heart Rate | 30 days of assigned diet
  Heart Rate will be determined in beats per minute using an automated blood pressure cuff following a 10 minute rest.
Resting Heart Rate | 60 days of assigned diet
  Heart Rate will be determined in beats per minute using an automated blood pressure cuff following a 10 minute rest.
Diastolic Blood Pressure | 0 days of assigned diet (baseline)
  Diastolic Blood Pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Diastolic Blood Pressure | 30 days of assigned diet
  Diastolic blood pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Diastolic Blood Pressure | 60 days of assigned diet
  Diastolic blood pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Systolic Blood Pressure | 0 days of assigned diet (baseline)
  Systolic blood pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Systolic Blood Pressure | 30 days of assigned diet
  Systolic blood pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Systolic Blood Pressure | 60 days of assigned diet
  Systolic blood pressure will be determined in millimeters mercury using an automated blood pressure cuff following a 10 minute rest.
Perceived wellness | 0 days of assigned diet (baseline)
  Perceived wellness will be self-reported using a 100 millimeter visual analog scale from 0 (very low) to 10 (extremely high) for self-esteem, energy level, motivation, irritability, focus, hunger, endurance, life satisfaction, physical appearance, and strength
Perceived wellness | 30 days of assigned diet
  Perceived wellness will be self-reported using a 100 millimeter visual analog scale from 0 (very low) to 10 (extremely high) for self-esteem, energy level, motivation, irritability, focus, hunger, endurance, life satisfaction, physical appearance, and strength
Perceived wellness | 60 days of assigned diet
  Perceived wellness will be self-reported using a 100 millimeter visual analog scale from 0 (very low) to 10 (extremely high) for self-esteem, energy level, motivation, irritability, focus, hunger, endurance, life satisfaction, physical appearance, and strength

OTHER OUTCOMES:
Digital images | 0 days of assigned diet (baseline)
  Digital images, for subjects consenting to photographing, will be collected from the subject's neck to knees from front, side, and back wearing form fitting clothing.
Digital images | 30 days of assigned diet
  Digital images, for subjects consenting to photographing, will be collected from the subject's neck to knees from front, side, and back wearing form fitting clothing.
Digital images | 60 days of assigned diet
  Digital images, for subjects consenting to photographing, will be collected from the subject's neck to knees from front, side, and back wearing form fitting clothing.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Stockton, PhD, Principal Investigator — University of Memphis
Locations (1):
- Center for Nutraceutical and Dietary Supplement Reseach, Memphis, Tennessee, United States